CLINICAL TRIAL: NCT04091412
Title: Study of Collateral Circulation and Related Gene Polymorphism in Patients With Symptomatic Intracranial Anterior Circulation Aortic Occlusion
Brief Title: Study of Collateral Circulation in Patients With Symptomatic Intracranial Anterior Circulation Occlusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, liuxiaoyun, Deputy Director of Neurology Department, The Second Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-P012
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Collateral Circulation; Large-artery Occlusion; Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long-term administration of Butylphthalide Soft Capsules (Experimental): In addition to standard secondary preventive drugs, such as atorvastatin calcium tablets, aspirin enteric-coated tablets and/or clopidogrel hydrogen sulphate tablets, patients in this group take Butylphthalide Soft Capsules orally, 0.2g per serving, three times a day for one year.
  Interventions: Drug: Butylphthalide Soft Capsules
- Standard secondary prevention group (No Intervention): patients in this group take atorvastatin calcium tablets, aspirin enteric-coated tablets and/or clopidogrel hydrogen sulphate tablets as standard secondary prevention.

INTERVENTIONS:
Drug: Butylphthalide Soft Capsules — The first class national new drug for the Treatment of Mild to Moderate Acute Ischemic Stroke; Long-term application can improve collateral circulation.
  Other Names: NBP
  Arms: Long-term administration of Butylphthalide Soft Capsules

SUMMARY:
Intracranial artery stenosis is the leading cause of stroke onset or recurrence in Asian. Multiple studies have shown that anterior circulation is most common in intracranial artery stenosis, especially the middle cerebral artery in patients with symptomatic or asymptomatic ischemic stroke. Based on the clinical experiences, we found that the cerebral collateral development can affect clinical symptoms seriously in patients with large artery stenosis. Compensated blood flow can reach the ischemic area through collateral circulation (including circle of Willis, leptomeningeal collaterals, extracranial to intracranial collaterals, and new angiogenesis) when the blood-supplying artery of the brain is severely stenotic or even occluded, however, considerable differences across individuals exist. Studies have shown statins and butylphthalide can promote collateral circulation. The influencing factors on collateral circulation building have not been completely identified yet, but a recent research found that Naturally occurring variants of Rabep2（Rab GTPase binding effector protein 2）are major determinants of variation in collateral extent and stroke severity in mice. On this basis, clinical trials have been conducted in order to confirm that the Rabep2 gene is associated with individual differences in the collateral circulation.

Summarizing new findings, we suspect whether the difference in the degree of collateral circulation is significant for long-term prognosis in patients with cerebral large arterial occlusion, and whether promoting collateral circulation and new angiogenesis can become a new treatment approach. Hereby, we plan to recruit 500 patients with cerebral large-artery occlusion, collect clinical and Imaging (CTA) information, analyze and investigate if the difference in the degree of collateral circulation can be the independent influencing factor for long-term prognosis. This study will collect blood sample of patients and further examine SNPs of Rabep2, and will then analyze the correlation between Rabep2 and patients with cerebral large-artery occlusion. This project will follow up rolled patients for 1 year, observe if long-term intake of butylphthalide can promote cerebral collateral development.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with arterial occlusion on unilateral or bilateral intracranial segment of internal carotid artery and/or middle cerebral artery were diagnosed by CTA; 2 complete medical records;

Exclusion Criteria:

1. CTA showed no arterial occlusion on unilateral or bilateral intracranial segment of internal carotid artery and/or middle cerebral artery; 2. Follow-up interventional surgery; 3. Death within 30 days of onset; 4. Clinical data incomplete; 5. Loss of follow-up patient.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
collateral circulation level | 1 hour
  Evaluation of collateral circulation level based on CTA

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Liu, Prf., Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- Second hospital of hebei medical university, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Zhang K, Liu L, Li T, Wang R, Bu K, Zhao P, Liu X. Collateral Circulation and Rabep2 Polymorphisms in Large Artery Occlusion: Impacts on Short- and Long-Term Prognosis. J Am Heart Assoc. 2025 Apr 15;14(8):e040032. doi: 10.1161/JAHA.124.040032. Epub 2025 Apr 10. PMID 40207533